CLINICAL TRIAL: NCT02829346
Title: Peri-articular Tranexamic Acid Injection in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Peri-articular Tranexamic Acid Injection in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, piya pinsornsak, Dr., Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-OT-0-096/54
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Tranexamic acid; Peri-articular injection; Total knee arthroplasty; Blood loss; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peri-articular group (Experimental): Patients received 750 mg of peri-articular Tranexamic acid (Transamin®; OLIC Thailand Ltd, Bangkok, Thailand; 250 mg/5 mL, 15 cc total volume) injection into the soft tissue around medial capsule (5 ml), lateral capsule (5 ml) and around the quadriceps muscle (5 ml), 10 minutes prior to deflating the tourniquet and wound closure.
  Interventions: Drug: Peri-articular tranexamic acid
- Intravenous group (Active Comparator): Patients received 750 mg of intravenous tranexamic acid(250 mg/5 ml, 15 cc total volume, keeping within the therapeutic range of 10-15 mg/kg/dose), 10 minutes prior to deflating the tourniquet and wound closure.
  Interventions: Drug: Intravenous tranexamic acid

INTERVENTIONS:
Drug: Peri-articular tranexamic acid — 750 mg of peri-articular TXA, prior to deflating the tourniquet and wound closure
  Other Names: Transamin
  Arms: Peri-articular group
Drug: Intravenous tranexamic acid — 750 mg of IV TXA, prior to deflating the tourniquet and wound closure
  Other Names: Transamin
  Arms: Intravenous group

SUMMARY:
This study evaluates the peri-articular tranexamic acid injection in total knee arthroplasty which is an alternative route of administration for blood loss reduction. Half of participants will receive intravenous tranexamic acid injection, while the other half will receive peri-articular tranexamic acid injection during total knee arthroplasty.

DETAILED DESCRIPTION:
Intravenous tranexamic acid (IV TXA) is one of the most effective agents in use for reducing blood loss following total knee arthroplasty (TKA) but its safety regarding venous thromboembolic events (VTEs) remains in question. The direct, local application of TXA may reduce systemic toxicity whilst maintaining good or better bleeding control compared to IV TXA. The topical application of TXA via Hemovac drains has been reported previously with good results. However, there are no data on peri-articular TXA injections during TKA.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with osteoarthritis in need of a TKA

Exclusion Criteria:

* inflammatory arthritis
* post-traumatic arthritis
* a history of or current venous thromboembolic disease
* any underlying disease of haemostasis
* cirrhosis
* chronic renal failure
* patients on anticoagulants or strong antiplatelet drugs (e.g. warfarin, clopidogrel)
* know allergy to TXA
* defective color vision
* preoperative hemoglobin <10 g/dL
* platelet count < 140,000 /uL3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The volume of postoperative blood loss in the drain | 48 hours after the operation
Changes from baseline hemoglobin concentrations | 48 hours after the operation
unit of blood transfusion | 48 hours after the operation

SECONDARY OUTCOMES:
Knee diameter for swelling | At 24 and 48 hours after the operation
number of patient with venous thromboembolism | At 14 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Piya Pinsornsak, MD, Principal Investigator — Faculty of Medicine, Thammasat university
Locations (1):
- Orthopaedic department, Thammasat university hospital, Klongluang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinclair KC, Clarke HD, Noble BN. Blood management in total knee arthroplasty: a comparison of techniques. Orthopedics. 2009 Jan;32(1):19. doi: 10.3928/01477447-20090101-21. PMID 19226044
- [Background] Gonzalez-Porras JR, Colado E, Conde MP, Lopez T, Nieto MJ, Corral M. An individualized pre-operative blood saving protocol can increase pre-operative haemoglobin levels and reduce the need for transfusion in elective total hip or knee arthroplasty. Transfus Med. 2009 Feb;19(1):35-42. doi: 10.1111/j.1365-3148.2009.00908.x. PMID 19302453
- [Background] Parvizi J, Diaz-Ledezma C. Total knee replacement with the use of a tourniquet: more pros than cons. Bone Joint J. 2013 Nov;95-B(11 Suppl A):133-4. doi: 10.1302/0301-620X.95B11.32903. PMID 24187371
- [Background] Sabatini L, Trecci A, Imarisio D, Uslenghi MD, Bianco G, Scagnelli R. Fibrin tissue adhesive reduces postoperative blood loss in total knee arthroplasty. J Orthop Traumatol. 2012 Sep;13(3):145-51. doi: 10.1007/s10195-012-0198-7. Epub 2012 May 16. PMID 22588333
- [Background] Pitta M, Zawadsky M, Verstraete R, Rubinstein A. Intravenous administration of tranexamic acid effectively reduces blood loss in primary total knee arthroplasty in a 610-patient consecutive case series. Transfusion. 2016 Feb;56(2):466-71. doi: 10.1111/trf.13354. Epub 2015 Oct 28. PMID 26509250
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Aggarwal AK, Singh N, Sudesh P. Topical vs Intravenous Tranexamic Acid in Reducing Blood Loss After Bilateral Total Knee Arthroplasty: A Prospective Study. J Arthroplasty. 2016 Jul;31(7):1442-8. doi: 10.1016/j.arth.2015.12.033. Epub 2015 Dec 21. PMID 26947543
- [Background] Benoni G, Lethagen S, Fredin H. The effect of tranexamic acid on local and plasma fibrinolysis during total knee arthroplasty. Thromb Res. 1997 Feb 1;85(3):195-206. doi: 10.1016/s0049-3848(97)00004-2. PMID 9058494
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Eubanks JD. Antifibrinolytics in major orthopaedic surgery. J Am Acad Orthop Surg. 2010 Mar;18(3):132-8. PMID 20190103
- [Background] Kluft C, Verheijen JH, Jie AF, Rijken DC, Preston FE, Sue-Ling HM, Jespersen J, Aasen AO. The postoperative fibrinolytic shutdown: a rapidly reverting acute phase pattern for the fast-acting inhibitor of tissue-type plasminogen activator after trauma. Scand J Clin Lab Invest. 1985 Nov;45(7):605-10. doi: 10.3109/00365518509155267. PMID 3934744
- [Background] Murphy WG, Davies MJ, Eduardo A. The haemostatic response to surgery and trauma. Br J Anaesth. 1993 Feb;70(2):205-13. doi: 10.1093/bja/70.2.205. No abstract available. PMID 7679584
- [Background] Charoencholvanich K, Siriwattanasakul P. Tranexamic acid reduces blood loss and blood transfusion after TKA: a prospective randomized controlled trial. Clin Orthop Relat Res. 2011 Oct;469(10):2874-80. doi: 10.1007/s11999-011-1874-2. Epub 2011 Apr 22. PMID 21512813
- [Background] Orpen NM, Little C, Walker G, Crawfurd EJ. Tranexamic acid reduces early post-operative blood loss after total knee arthroplasty: a prospective randomised controlled trial of 29 patients. Knee. 2006 Mar;13(2):106-10. doi: 10.1016/j.knee.2005.11.001. Epub 2006 Feb 17. PMID 16487712
- [Background] Ortega-Andreu M, Perez-Chrzanowska H, Figueredo R, Gomez-Barrena E. Blood loss control with two doses of tranexamic Acid in a multimodal protocol for total knee arthroplasty. Open Orthop J. 2011 Mar 16;5:44-8. doi: 10.2174/1874325001105010044. PMID 21552468
- [Background] Mannucci PM. Hemostatic drugs. N Engl J Med. 1998 Jul 23;339(4):245-53. doi: 10.1056/NEJM199807233390407. No abstract available. PMID 9673304
- [Background] Mannucci PM, Levi M. Prevention and treatment of major blood loss. N Engl J Med. 2007 May 31;356(22):2301-11. doi: 10.1056/NEJMra067742. No abstract available. PMID 17538089
- [Background] Ishida K, Tsumura N, Kitagawa A, Hamamura S, Fukuda K, Dogaki Y, Kubo S, Matsumoto T, Matsushita T, Chin T, Iguchi T, Kurosaka M, Kuroda R. Intra-articular injection of tranexamic acid reduces not only blood loss but also knee joint swelling after total knee arthroplasty. Int Orthop. 2011 Nov;35(11):1639-45. doi: 10.1007/s00264-010-1205-3. Epub 2011 Jan 21. PMID 21253725
- [Background] Maniar RN, Kumar G, Singhi T, Nayak RM, Maniar PR. Most effective regimen of tranexamic acid in knee arthroplasty: a prospective randomized controlled study in 240 patients. Clin Orthop Relat Res. 2012 Sep;470(9):2605-12. doi: 10.1007/s11999-012-2310-y. Epub 2012 Mar 15. PMID 22419350
- [Background] Roy SP, Tanki UF, Dutta A, Jain SK, Nagi ON. Efficacy of intra-articular tranexamic acid in blood loss reduction following primary unilateral total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2012 Dec;20(12):2494-501. doi: 10.1007/s00167-012-1942-5. Epub 2012 Mar 15. PMID 22419263
- [Background] Wang H, Shen B, Zeng Y. Blood Loss and Transfusion After Topical Tranexamic Acid Administration in Primary Total Knee Arthroplasty. Orthopedics. 2015 Nov;38(11):e1007-16. doi: 10.3928/01477447-20151020-10. PMID 26558665
- [Background] Spreng UJ, Dahl V, Hjall A, Fagerland MW, Raeder J. High-volume local infiltration analgesia combined with intravenous or local ketorolac+morphine compared with epidural analgesia after total knee arthroplasty. Br J Anaesth. 2010 Nov;105(5):675-82. doi: 10.1093/bja/aeq232. Epub 2010 Aug 24. PMID 20736233
- [Background] Manor D, Sadeh M. Muscle fibre necrosis induced by intramuscular injection of drugs. Br J Exp Pathol. 1989 Aug;70(4):457-62. PMID 2765397
- [Background] Pinsornsak P, Chumchuen S. Can a modified Robert Jones bandage after knee arthroplasty reduce blood loss? A prospective randomized controlled trial. Clin Orthop Relat Res. 2013 May;471(5):1677-81. doi: 10.1007/s11999-013-2786-0. Epub 2013 Jan 11. PMID 23307631
- [Background] Kagoma YK, Crowther MA, Douketis J, Bhandari M, Eikelboom J, Lim W. Use of antifibrinolytic therapy to reduce transfusion in patients undergoing orthopedic surgery: a systematic review of randomized trials. Thromb Res. 2009 Mar;123(5):687-96. doi: 10.1016/j.thromres.2008.09.015. Epub 2008 Nov 12. PMID 19007970
- [Background] Alshryda S, Sarda P, Sukeik M, Nargol A, Blenkinsopp J, Mason JM. Tranexamic acid in total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Br. 2011 Dec;93(12):1577-85. doi: 10.1302/0301-620X.93B12.26989. PMID 22161917
- [Derived] Pinsornsak P, Rojanavijitkul S, Chumchuen S. Peri-articular tranexamic acid injection in total knee arthroplasty: a randomized controlled trial. BMC Musculoskelet Disord. 2016 Jul 26;17:313. doi: 10.1186/s12891-016-1176-7. PMID 27455842